CLINICAL TRIAL: NCT00357851
Title: Can Aprotinin Reduce Pancreatitis After Scoliosis Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: IRB#2003-029
Record Dates: First submitted 2006-07-26; First posted 2006-07-28 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-10

CONDITIONS: Pancreatitis
Keywords: pancreatitis, blood loss
MeSH Terms: conditions — Pancreatitis; Hemorrhage | interventions — Aprotinin

INTERVENTIONS:
Drug: Aprotinin

SUMMARY:
Pancreatitis is caused by an acute injury on the pancreas. This illness is associated with abdominal pain, vomiting or even fever. We have recently reported a high rate of acute pancreatitis developing in children who undergo posterior spinal fusion for scoliosis (to correct spinal curve). We showed that the amount of blood loss during the surgery is related to the incidence of pancreatitis. In addition, some markers that monitor tissue injury are elevated after the surgery and significantly higher in the patients who develop acute pancreatitis later. We propose that if blood loss and tissue injury could be reduced, then the incidence of pancreatits may be less in these children. Therefore we plan to use a drug Aprotinin to just do that. Aprotinin has been used to reduce blood loss in patients undergoing posterior spinal surgery, the same population we propose to study. If it turns out that Aprotinin can reduce blood loss or/and the damage to the pancreas, thus pancreatitis, it will diminish the pain and discomfort, and shorten hospital stay in these children. The results from this study will guide medical care in these children in the future.

DETAILED DESCRIPTION:
We have shown an association between high intraoperative blood loss in children and young adults undergoing posterior spinal fusion and a subsequent clinical course characterized by a high rate of acute pancreatitis - a rare illness in children. Other complications include sepsis, deep wound infections, and prolonged length of stay. Although it has been reported in children and young adults with idiopathic scoliosis we have shown a significantly higher blood loss and rate of pancreatitis in patients with neuromuscular scoliosis, especially in cerebral palsy. The purpose of this study is to assess the efficacy of Aprotinin, a serine protease inhibitor, in reducing intraoperative blood loss and subsequent clinical pancreatitis and other associated complications in patients with cerebral palsy who undergo posterior spinal fusion. Aprotinin is currently approved for use in adults to reduce major blood loss during cardiac surgery, and it is used in children at virtually all major pediatric cardiac centers. In these populations, blood loss is consistently diminished by 50%. Safety and efficacy in adults and children is well documented, and use of this drug is familiar to most anesthesiologists. In addition, it has been shown to reduce blood loss effectively in large controlled-studies in adults who undergo major orthopedic surgeries, including spinal fusion. Recently one published study has also suggested that Aprotinin may reduced blood loss in children undergoing idiopathic scoliosis surgery, but the study did not have the adequately statistical power due to a small sample size. Since intraoperative blood loss and cytokine elevations are significantly correlated with the incidence of acute pancreatitis, we hypothesize a major role for ischemic injury in the development of pancreatitis and other complications. We expect that Aprotinin by reducing blood loss will prevent ischemic injury hence, decrease the incidence of acute pancreatitis in these children and young adults. While safety and efficacy have been established for cardiac surgery in adults and children, we propose to conduct a double-blind, randomized trial of Aprotinin in children with cerebral palsy who undergo posterior spinal fusion surgery to answer the following specific questions.

Specific Aim 1: To assess whether intraoperative Aprotinin infusion can reduce intraoperative blood loss, and whether this lowers the incidence of postoperative pancreatitis and associated complications of sepsis, wound infection and prolonged length of stay.

Specific Aim 2: To assess by indirect methods whether Aprotinin infusion can alter the degree of ischemic injury concomitantly with the reduction of blood loss and the incidence of postoperative pancreatitis.

ELIGIBILITY:
Inclusion Criteria:

Children of all ages (<18 yr or 18 yr), both boys and girls who undergo posterior spinal fusion with cebebral palsy or neuromuscular scoliosis.

Exclusion Criteria:

* received Aprotinin previously
* have severe allergic reaction to medicine
* received whole blood transfusions
* bleeding disorder
* impaired renal function, liver or kidney impairment
* previous pancreatitis
* girls who are pregnant.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-03

PRIMARY OUTCOMES:
Blood loss and the incidence of pancreatitis

SECONDARY OUTCOMES:
Ischemic injury

CONTACTS AND LOCATIONS:
Locations (1):
- Alfred I. duPont Hospital for Children, Wilmington, Delaware, United States